CLINICAL TRIAL: NCT03759873
Title: Improving Participation in Cardiac Rehabilitation Among Lower-Socioeconomic Status Patients: Efficacy of Early Case Management and Financial Incentives
Brief Title: Incentives and Case Management to Improve Cardiac Care: Healthy Lifestyle Program
Acronym: HeLP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Diann Gaalema, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R61HL143305 (NIH)
Record Dates: First submitted 2018-11-20; First posted 2018-11-30 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Rehabilitation
Keywords: Incentives; Case management; Socioeconomic status
MeSH Terms: interventions — Fertility; Case Management

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Incentives (Experimental): Patient earns incentives for completing cardiac rehabilitation sessions.
  Interventions: Behavioral: Incentives
- Case Management (Experimental): Patient is assigned a case manager while in hospital.
  Interventions: Behavioral: Case Management
- Incentives and Case Management (Experimental): Patient receives both the Incentives and Case Management interventions.
  Interventions: Behavioral: Incentives; Behavioral: Case Management
- Usual care (No Intervention): This control condition does not receive either intervention.

INTERVENTIONS:
Behavioral: Incentives — Patient earns financial incentives (gift cards) on an escalating schedule for completing cardiac rehabilitation sessions.
  Arms: Incentives; Incentives and Case Management
Behavioral: Case Management — A case manager is available by phone to assist patient with attending cardiac rehabilitation sessions as well as to provide advice about cardiac symptoms and healthy behavior change.
  Arms: Case Management; Incentives and Case Management

SUMMARY:
Participation in outpatient cardiac rehabilitation (CR) decreases morbidity and mortality for patients hospitalized with myocardial infarction, coronary bypass surgery or percutaneous revascularization. Unfortunately, only 10-35% of patients for whom CR is indicated choose to participate. Lower socioeconomic status (SES) is a robust predictor of CR non-participation. There is growing recognition of the need to increase CR among economically disadvantaged patients, but there are almost no evidence-based interventions available for doing so. The present study will examine the efficacy of using early case management and financial incentives for increasing CR participation among lower-SES patients. Case management has been effective at promoting attendance at a variety of health-related programs (e.g. treatment for diabetes, HIV, asthma, cocaine dependence) as well as reducing hospitalizations. Financial incentives are also highly effective in altering health behaviors among disadvantaged populations (e.g., smoking during pregnancy, weight loss) including CR participation in a prior trial. For this study 209 CR-eligible lower-SES patients will be randomized to: a treatment condition where patients are assigned a case manager while in hospital who will facilitate CR attendance and coordinate cardiac care, a treatment condition where patients receive financial incentives contingent on initiation of and continued attendance at CR sessions, a combination of these two interventions, or to a "usual-care" condition. Participants in all conditions will complete pre- and post-treatment assessments. Treatment conditions will be compared on attendance at CR and end-of-intervention improvements in fitness, executive function, and health-related quality of life. Cost effectiveness of the treatment conditions will also be examined by comparing the costs of delivering the interventions and the usual care condition, taking into account increases in CR participation. Furthermore, the value of the interventions will be modeled based on increases in participation rates, intervention costs, long-term medical costs, and health outcomes after a coronary event. This systematic examination of promising interventions will allow testing of the efficacy and cost-effectiveness of approaches that have the potential to substantially increase CR participation and significantly improve health outcomes among lower-SES cardiac patients.

ELIGIBILITY:
Inclusion Criteria:

* A recent myocardial infarction, coronary revascularization, diagnosis of congestive heart failure (CHF) or heart valve replacement or repair
* Enrolled in a state-supported insurance plan for low income individuals or receiving other state benefits that are based on financial need (housing subsidy, food stamps, etc.), or with a less than high school education.
* Lives in and plans to remain in the greater Burlington, Vermont area (Chittenden county) for the next 12 mos.
* Copley Hospital (Morrisville, VT) transfer patient (enrolled in a state-supported insurance plan for low income individuals or receiving other state benefits that are based on financial need)
* Northwestern Medical Center (St Albans, VT) transfer patient (enrolled in a state-supported insurance plan for low income individuals or receiving other state benefits that are based on financial need)

Exclusion Criteria:

* Dementia (MMSE<20) or current untreated Axis 1 psychiatric disorder other than nicotine dependence as determined by medical history
* Advanced cancer, advanced frailty, or other longevity-limiting systemic disease that would preclude CR participation
* Rest angina or very low threshold angina (<2 METS) until adequate therapy is instituted
* Severe life threatening ventricular arrhythmias unless adequately controlled (e.g. intracardiac defibrillator)
* Class 4 chronic heart failure (symptoms at rest)
* Exercise-limiting non-cardiac disease such as severe arthritis, past stroke, severe lung disease
* Previous successful attendance at cardiac rehabilitation (defined as completing 6+ sessions in the past 10 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaalema DE, Khadanga S, Savage PD, Yant B, Katz BR, DeSarno M, Ades PA. Improving Cardiac Rehabilitation Adherence in Patients With Lower Socioeconomic Status: A Randomized Clinical Trial. JAMA Intern Med. 2024 Sep 1;184(9):1095-1104. doi: 10.1001/jamainternmed.2024.3338. PMID 39037811

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Started | 57 | 57 | 57 | 38
Completed | 53 | 51 | 52 | 36
Not Completed | 4 | 6 | 5 | 2
Not completed — Not appropriate for cardiac rehab | 4 | 4 | 4 | 2
Not completed — Moved outside eligible area | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care | Total
Number analyzed (Participants) | 53 | 51 | 52 | 36 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 42 | 27 | 147
  >=65 years | 14 | 12 | 10 | 9 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.2) | 57.9 (12.7) | 57.9 (10.9) | 57.1 (10.5) | 57.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 21 | 20 | 14 | 67
  Male | 41 | 30 | 32 | 22 | 125
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic White | 0 | 3 | 0 | 0 | 3
  Hispanic Other/Multiracial | 1 | 0 | 0 | 0 | 1
  Black or African American | 3 | 4 | 1 | 1 | 9
  Asian | 1 | 0 | 0 | 2 | 3
  American Indian | 2 | 1 | 1 | 1 | 5
  Other/Multiracial | 2 | 2 | 2 | 3 | 9
  Non-Hispanic White | 44 | 41 | 48 | 29 | 162
Region of Enrollment [Number; unit: participants]
  United States | 53 | 51 | 52 | 36 | 192
Primary Diagnosis [Count of Participants; unit: Participants]
  Percutaneous Intervention | 27 | 27 | 31 | 23 | 108
  Coronary Artery Bypass Graft | 12 | 7 | 6 | 4 | 29
  Valve Replacement/Repair | 7 | 8 | 5 | 2 | 22
  Chronic Systolic Heart Failure | 6 | 6 | 4 | 5 | 21
  Myocardial Infarction | 1 | 1 | 5 | 2 | 9
  Stable Angina | 0 | 2 | 1 | 0 | 3
Currently Smoking [Count of Participants; unit: Participants] | 23 | 21 | 23 | 18 | 85
Patient Health Questionnaire-2 [Count of Participants; unit: Participants]
  Screen Negative (0-2) | 39 | 41 | 40 | 25 | 145
  Screen Positive (0-2) | 13 | 10 | 11 | 11 | 45
  Data Missing | 1 | 0 | 1 | 0 | 2
Enrolled in Medicaid [Count of Participants; unit: Participants] | 52 | 48 | 50 | 35 | 185
Education [Count of Participants; unit: Participants]
  Less Than High School/GED | 11 | 19 | 8 | 11 | 49
  High School/Some College | 28 | 22 | 28 | 15 | 93
  College/Advanced Degree | 13 | 10 | 16 | 10 | 49
  Data Missing | 1 | 0 | 0 | 0 | 1
Region [Count of Participants; unit: Participants]
  Rural | 16 | 14 | 15 | 3 | 48
  Urban | 37 | 37 | 37 | 33 | 144
Peak Oxygen Uptake (Peak VO2) [Mean (Standard Deviation); unit: milliliters per kilogram per minute] | 17.9 (6.3) | 16.8 (5.5) | 18.8 (5.5) | 17.7 (6.7) | 17.9 (5.9)
Estimated Metabolic Equivalent of Task (METs) [Mean (Standard Deviation); unit: kilocalories per kilogram per hour] | 5.8 (2.7) | 5.5 (2.3) | 6.2 (2.2) | 6.4 (3.0) | 5.9 (2.5)
Waist Circumference [Mean (Standard Deviation); unit: inches] | 41.3 (6.4) | 44.6 (8.7) | 43.0 (6.8) | 42.2 (6.3) | 42.8 (7.2)
Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — Depressive symptoms at baseline will be measured using the "The Beck Depression Inventory (BDI)." Scores range from 0 to 63, with higher scores indicating worse outcomes.
  units on a scale | 9.3 (7.5) | 14.6 (10.4) | 11.1 (8.2) | 17.5 (13.7) | 12.6 (10.0)
MacNew Heart Disease Health-related Quality of Life Questionnaire [Least Squares Mean (Standard Deviation); unit: units on a scale] — Perceived quality of life will be measured at intake using the MacNew Heart Disease Health-Related Quality of Life Questionnaire. Scores range from 1 to 7, with higher scores indicating better outcomes.
  units on a scale | 5.0 (1.0) | 4.9 (1.1) | 5.1 (1.0) | 4.7 (1.3) | 4.9 (1.1)
EuroQol Visual Analogue Scale [Mean (Standard Deviation); unit: units on a scale] — Perceived quality of life at intake will be measured using the Visual Analogue Scale of the EuroQol-5D-3L. Scores range from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 64.1 (16.4) | 55.2 (22.4) | 60.1 (19.3) | 62.4 (20.9) | 60.2 (19.9)

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Rehabilitation Attendance
Description: Number of cardiac rehabilitation sessions completed out of a possible 36
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: sessions of CR
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
sessions of CR | 16.9 [12.7 to 21.1] | 12.0 [7.7 to 16.1] | 24.1 [19.9 to 28.4] | 10.9 [5.8 to 15.9]

2. Primary Outcome: Cardiac Rehabilitation Completion
Description: Proportion of patients who complete 30+ sessions of cardiac rehabilitation
Time Frame: Within 4 months of the intake assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
Participants | 22 | 13 | 32 | 4

3. Secondary Outcome: Change in Fitness (Peak Oxygen Uptake)
Description: Changes in fitness level (peak oxygen uptake) will be measured from intake to completion of the intervention (4 months after intake).
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters per kilogram per minute
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
milliliters per kilogram per minute | 20.9 [20.0 to 21.9] | 18.3 [17.3 to 19.3] | 18.6 [17.7 to 19.5] | 21.2 [19.8 to 22.6]

4. Secondary Outcome: Change in Fitness (Estimated Metabolic Equivalent of Task)
Description: Changes in fitness level (Metabolic Equivalent of Tasks) will be measured from intake to completion of the intervention (4 months after intake).
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters per kilogram per minute
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
milliliters per kilogram per minute | 7.4 [6.8 to 8.1] | 6.5 [5.8 to 7.2] | 7.0 [6.3 to 7.7] | 6.7 [5.7 to 7.8]

5. Secondary Outcome: Change in Body Composition
Description: Changes in waist measurement will be measured from intake to completion of the intervention (4 months after intake).
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: inches
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
inches | 42.1 [41.6 to 42.6] | 42.7 [42.1 to 43.2] | 42.1 [41.7 to 42.6] | 42.0 [41.3 to 42.7]

6. Secondary Outcome: Changes in Smoking Status
Description: Changes in smoking status will be measured from intake to completion of the intervention (4 months after intake).
Time Frame: Within 4 months of the intake assessment
Population: Overall number of participants analyzed represents the total number of participants from each arm of the study who completed this measure and for whom data were collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 30 | 28 | 39 | 17
Participants | 8 | 10 | 11 | 5

7. Secondary Outcome: Changes in Quality of Life - Cardiac Specific
Description: Changes in perceived quality of life (MacNew) questionnaires will be measured from intake to completion of the intervention (4 months after intake). The MacNew Heart Disease Health-Related Quality of Life Questionnaire was used. Scores range from 1 to 7, with higher scores indicating better outcomes.
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
score on a scale | 5.4 [5.3 to 5.6] | 5.4 [5.2 to 5.6] | 5.2 [5.1 to 5.4] | 5.4 [5.2 to 5.7]

8. Secondary Outcome: Changes in Quality of Life - Non-specific
Description: Changes in perceived quality of life (EuroQoL) questionnaires will be measured from intake to completion of the intervention (4 months after intake). The Visual Analogue Scale of the EuroQol-5D-3L was used. Scores range from 0 to 100, with higher scores indicating better outcomes.
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
score on a scale | 66.0 [61.9 to 70.2] | 66.2 [61.5 to 70.9] | 70.3 [66.2 to 74.3] | 64.0 [57.7 to 70.4]

9. Secondary Outcome: Changes in Mental Health
Description: Changes in mental health (Adult Self-Report) questionnaires will be measured from intake to completion of the intervention (4 months after intake) using the Achenbach System of Empirically Based Assessment (ASEBA). T-scores are reported. A T-score of 50 indicates the population mean, and 10 is the standard deviation. Higher T-scores indicate worse outcomes. T-scores above 63 indicate clinically significant problems, and those between 60 and 63 fall within the borderline clinical range.
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: T scores
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
T scores | 54.16 [52.45 to 55.86] | 55.58 [53.70 to 57.46] | 55.41 [53.86 to 56.96] | 52.82 [50.33 to 55.31]

10. Secondary Outcome: Changes in Depressive Symptoms
Description: Changes in reported depressive symptoms "The Beck Depression Inventory (BDI)" will be measured from intake to completion of the intervention (4 months after intake). BDI results will be back transformed due to data being square root transformed. Scores range from 0 to 63, with higher scores indicating worse outcomes.
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
score on a scale | 9.0 [7.3 to 10.8] | 6.6 [5.1 to 8.3] | 9.1 [7.5 to 10.9] | 6.6 [4.7 to 8.8]

11. Secondary Outcome: Changes in Executive Function (Delay Discounting)
Description: Changes in Executive function (delay discounting) will be measured from intake to completion of the intervention (4 months after intake). A 5-trial adjusting delay discounting task was used to calculate k values, numerical representations of the rate of discounting. k values range from 0 to 0.5, with larger values indicating steeper discounting (more impulsivity; greater propensity to devalue delayed rewards in favor of more immediate outcomes). k values were log(10) transformed for analysis. Larger log transformed k values indicate steeper discounting.
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: log of k
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
log of k | -1.82 [-2.11 to -1.52] | -1.94 [-2.26 to -1.61] | -2.32 [-2.58 to -2.05] | -2.52 [-2.91 to -2.13]

12. Secondary Outcome: Changes in Executive Function (DS)
Description: Changes in Executive function (digit span) will be measured from intake to completion of the intervention (4 months after intake). The Digit Span subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) was used. Scores range from 1 to 19, with higher scores indicating worse outcomes.
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
score on a scale | 8.51 [8.13 to 8.90] | 8.21 [7.77 to 8.65] | 9.16 [8.82 to 9.51] | 8.87 [8.35 to 9.39]

13. Secondary Outcome: Changes in Executive Function (Trail)
Description: Changes in Executive function (Trail making task) will be measured from intake to completion of the intervention (4 months after intake). The Trail-Making subtest of the Delis-Kaplan Executive Function System (D-KEFS) was used. Scores range from 1 to 19, with higher scores indicating worse outcomes.
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
score on a scale | 10.19 [9.59 to 10.78] | 10.19 [9.46 to 10.93] | 10.29 [9.74 to 10.85] | 11.01 [10.22 to 11.80]

14. Secondary Outcome: Changes in Executive Function (BRIEF)
Description: Changes in self-reported Executive function problems (BRIEF) will be measured from intake to completion of the intervention (4 months after intake). The Global Executive Composite (GEC) of the Behavior Rating Inventory of Executive Function (BRIEF) was used. T-scores are reported. A T-score of 50 indicates the population mean, and 10 is the standard deviation. Higher T-scores indicate worse outcomes. T-scores above 65 indicate clinically significant problems.
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: T scores
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
T scores | 55.35 [53.54 to 57.15] | 56.64 [54.44 to 58.84] | 55.67 [53.96 to 57.39] | 54.91 [52.43 to 57.39]

15. Secondary Outcome: Changes in Executive Function (SST)
Description: Changes in Executive function (Stop Signal Task) will be measured from intake to completion of the intervention (4 months after intake).
Time Frame: Within 4 months of the intake assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
seconds | 180.86 [162.62 to 199.09] | 182.53 [163.40 to 201.65] | 221.77 [206.75 to 236.80] | 165.26 [141.26 to 189.26]

16. Secondary Outcome: Health Care Contacts
Description: Combined measure of number of Emergency Department (ED) visits and overnight hospitalizations.
Time Frame: One year period starting at intake assessment.
Measure: Number; unit: number of visits
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 53 | 51 | 52 | 36
number of visits | 113 | 180 | 201 | 142

17. Secondary Outcome: Health Care Costs
Description: Costs associated with combined Emergency Department (ED) visits and overnight hospitalizations.
Time Frame: One year period starting at intake assessment.
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Maintenance of Fitness Following Intervention (Peak Oxygen Uptake)
Description: Changes in fitness level (peak oxygen uptake) will be measured from intervention completion until follow-up (8 months after intervention completion).
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milliliters per kilogram per minute
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 19 | 15 | 27 | 13
milliliters per kilogram per minute | 20.2 (5.8) | 18.5 (6.3) | 21.3 (7.4) | 19.0 (7.4)

19. Other Pre Specified Outcome: Maintenance of Fitness Following Intervention (Estimated Metabolic Equivalent of Task)
Description: Changes in fitness level (Estimated Metabolic Equivalent of Task) will be measured from intervention completion until follow-up (8 months after intervention completion).
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milliliters per kilogram per minute
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 19 | 15 | 27 | 13
milliliters per kilogram per minute | 6.4 (3.3) | 6.8 (3.0) | 7.4 (3.5) | 6.4 (2.8)

20. Other Pre Specified Outcome: Maintenance of Waist Circumference Following Intervention.
Description: Changes in waist circumference will be measured from intervention completion until follow-up (8 months after intervention completion).
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 23 | 23 | 33 | 18
inches | 42.5 (7.1) | 44.2 (8.8) | 42.0 (7.0) | 42.2 (7.4)

21. Other Pre Specified Outcome: Maintenance of Smoking Status Following Intervention.
Description: Changes in smoking status will be measured from intervention completion until follow-up (8 months after intervention completion).
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
Number analyzed (Participants) | 24 | 23 | 34 | 18
Participants | 7 | 9 | 12 | 3

22. Other Pre Specified Outcome: Maintenance of Quality of Life (Cardiac-specific) Following Intervention.
Description: Changes in perceived quality of life (MacNew) questionnaires will be measured from intervention completion until follow-up (8 months after intervention completion). The MacNew Heart Disease Health-Related Quality of Life Questionnaire was used. Scores range from 1 to 7, with higher scores indicating better outcomes.
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Maintenance of Quality of Life (Noncardiac-specific) Following Intervention.
Description: Changes in perceived quality of life (EuroQoL) questionnaires will be measured from intervention completion until follow-up (8 months after intervention completion). The Visual Analogue Scale of the EuroQol-5D-3L was used. Scores range from 0 to 100, with higher scores indicating better outcomes.
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Maintenance of Mental Health Following Intervention.
Description: Changes in mental health (Adult Self-Report) questionnaires will be measured from intervention completion until follow-up (8 months after intervention completion) using the Achenbach System of Empirically Based Assessment (ASEBA). T-scores are reported. A T-score of 50 indicates the population mean, and 10 is the standard deviation. Higher T-scores indicate worse outcomes. T-scores above 63 indicate clinically significant problems, and those between 60 and 63 fall within the borderline clinical range.
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Maintenance of Depressive Symptoms Following Intervention.
Description: Changes in reported depressive symptoms "The Beck Depression Inventory (BDI)" will be measured from intervention completion until follow-up (8 months after intervention completion). BDI results will be back transformed due to data being square root transformed. Scores range from 0 to 63, with higher scores indicating worse outcomes.
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Maintenance of Executive Function (Delay Discounting) Following Intervention.
Description: Changes in Executive function (delay discounting) will be measured from intervention completion until follow-up (8 months after intervention completion). A 5-trial adjusting delay discounting task will be used to calculate k values, numerical representations of the rate of discounting. k values range from 0 to 0.5, with larger values indicating steeper discounting (more impulsivity; greater propensity to devalue delayed rewards in favor of more immediate outcomes). k values were log(10) transformed for analysis. Larger log transformed k values indicate steeper discounting.
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Maintenance of Executive Function (DS) Following Intervention.
Description: Changes in Executive function (digit span) will be measured from intervention completion until follow-up (8 months after intervention completion). The Digit Span subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) was used. Scores range from 1 to 19, with higher scores indicating worse outcomes.
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Maintenance of Executive Function (BRIEF) Following Intervention.
Description: Changes in self-reported Executive function problems (BRIEF) will be measured from intervention completion until follow-up (8 months after intervention completion). The Global Executive Composite (GEC) of the Behavior Rating Inventory of Executive Function (BRIEF) was used. T-scores are reported. A T-score of 50 indicates the population mean, and 10 is the standard deviation. Higher T-scores indicate worse outcomes. T-scores above 65 indicate clinically significant problems.
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Maintenance of Executive Function (SST) Following Intervention.
Description: Changes in Executive function (stop signal task) will be measured from intervention completion until follow-up (8 months after intervention completion).
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Maintenance of Executive Function (Trail) Following Intervention.
Description: Changes in Executive function (trail making task) will be measured from intervention completion until follow-up (8 months after intervention completion). The Trail-Making subtest of the Delis-Kaplan Executive Function System (D-KEFS) was used. Scores range from 1 to 19, with higher scores indicating worse outcomes.
Time Frame: From completion of intervention (4 months) to follow-up (one-year).
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Cost-effectiveness
Description: Cost-effectiveness of the intervention will be determined. Cost-effectiveness is a single outcome (cost per per quality-adjusted life year gained) that is calculated by integrating the cost of delivering the intervention, the cost to the patient of receiving the intervention, and the benefits both in quality of life and in reductions in healthcare utilization.
Time Frame: One year period starting at intake assessment.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 Year
Description: All participants were asked about their general health, symptoms, and adverse events once per week during scheduled weekly phone check-ins conducted by the study coordinator. Additionally, participants in the two case management arms had a second weekly check-in with their case manager during which they were asked about adverse events. Finally, the study team was notified via Epic whenever a participant was admitted to the hospital or ED.
Arm/Group | Incentives | Case Management | Incentives and Case Management | Usual Care
All-Cause Mortality (participants affected / at risk) | 3/53 | 5/51 | 3/52 | 0/36
Serious Adverse Events (participants affected / at risk) | 15/53 | 25/51 | 20/52 | 16/36
Other Adverse Events (participants affected / at risk) | 39/53 | 42/51 | 42/52 | 27/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incentives (N=53) | Case Management (N=51) | Incentives and Case Management (N=52) | Usual Care (N=36)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol Intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac Disorders - Other (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain - Cardiac (Cardiac disorders) | 2 (2) | 4 (5) | 5 (6) | 7 (10)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Colorectal Cancer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Bypass (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 3 (3) | 4 (4) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6) | 1 (1) | 3 (5)
Edema Limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to Thrive (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Gastric Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and Medical Procedures - Other (Surgical and medical procedures) | 4 (5) | 7 (8) | 2 (2) | 4 (4)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Thromboembolic Event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visceral Arterial Ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Wound Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incentives (N=53) | Case Management (N=51) | Incentives and Case Management (N=52) | Usual Care (N=36)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) | 7 (9)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 3 (3) | 4 (4)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 1 (1) | 4 (5) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 6 (8) | 9 (18) | 8 (16) | 7 (15)
Chest Pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colorectal cancer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Common Cold (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 4 (5)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dental abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Dizziness (Nervous system disorders) | 3 (4) | 2 (2) | 5 (7) | 1 (1)
Domestic violence assault (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (6) | 4 (4) | 6 (16)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Eye disorders - Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (5) | 5 (5) | 5 (5)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (5)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpes Simplex (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle cramp (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disord (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmares (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 3 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 8 (11) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 1 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disord (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Oth (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 2 (2) | 1 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 4 (5) | 7 (10) | 4 (5) | 6 (10)
Surgical and medical procedures - Other (Surgical and medical procedures) | 5 (6) | 3 (3) | 7 (11) | 4 (6)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urostomy leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision decreased (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound Treatment (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was powered for attendance rather than clinical outcomes; Study was conducted exclusively within Vermont, which may limit generalizability; Some assessment data are limited due to COVID-19 restrictions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03759873/Prot_SAP_004.pdf
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT03759873/ICF_003.pdf